CLINICAL TRIAL: NCT01585194
Title: Phase II Study of Nivolumab in Combination With Ipilimumab for Uveal Melanoma
Brief Title: Nivolumab and Ipilimumab in Treating Patients With Metastatic Uveal Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0919; NCI-2015-00853 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2012-00665; 2011-0919 (Other: M D Anderson Cancer Center); R21CA208609 (NIH)
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Uveal Melanoma; Stage IV Uveal Melanoma AJCC v7
MeSH Terms: conditions — Uveal Melanoma | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, ipilimumab) (Experimental): INDUCTION PHASE: Patients receive nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes during weeks 1, 4, 7, and 10. Treatment continues for 12 weeks in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Patients not experiencing disease progression or unacceptable toxicity by week 12 of the induction phase receive nivolumab IV every 2 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial studies how well nivolumab and ipilimumab work in treating patients with uveal melanoma that has spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Overall response rate.

SECONDARY OBJECTIVES:

I. Progression-free survival. II. Median overall survival. III. One-year overall survival.

EXPLORATORY OBJECTIVES:

I. Tissue and blood correlates to define immune infiltration and signatures as a result of treatment with nivolumab plus ipilimumab.

OUTLINE:

INDUCTION PHASE: Patients receive nivolumab intravenously (IV) over 60 minutes and ipilimumab IV over 90 minutes during weeks 1, 4, 7, and 10. Treatment continues for 12 weeks in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Patients not experiencing disease progression or unacceptable toxicity by week 12 of the induction phase receive nivolumab IV every 2 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* History of uveal melanoma and documented metastatic disease with at least one measurable lesion is required; which is >= 1 cm x 1 cm (on spiral computed tomography [CT] or equivalent)
* Any number of prior therapies is allowed
* White blood cell (WBC) >= 2000/uL
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelets >= 100 x 10^3/uL
* Hemoglobin >= 9 g/dL
* Creatinine =< 1.5 x upper limit of normal (ULN) or creatinine clearance (CrCl) > 40 mL/min (using the Cockcroft-Gault formula)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x ULN for patients without liver metastasis, =< 5 x ULN for liver metastases
* Bilirubin =< 1.5 x ULN, (except patients with Gilbert's syndrome, who must have a total bilirubin less than 3.0 mg/dL)
* In suspected patients no active or chronic infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-1
* Baseline imaging in the form of CT chest, abdomen, pelvis with oral and intravenous contrast within 28 days of study entry; for patients with a contrast allergy, choice of alternative body imaging will be at the discretion of the investigator or his designee; magnetic resonance imaging (MRI) of the brain is only needed if clinically indicated
* Prior to start of treatment must be more than 21 days elapsed from surgery, radiation therapy, or prior chemotherapy; more than 42 days elapsed from prior immune therapy including vaccines
* Women of childbearing potential (WOCBP) and fertile men with partners of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 26 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized

Exclusion Criteria:

* Untreated primary uveal melanoma except in cases where metastatic disease is diagnosed at the time of primary disease
* Metastatic uveal melanoma patients with bone-only disease
* Any other malignancy from which the patient has been disease-free for less than 2 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix, breast, or prostate
* Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]; motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis)
* Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of adverse events (AEs), such as a condition associated with frequent diarrhea
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab)
* Concomitant therapy with any of the following: tamoxifen, toremifene, IL 2, interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids greater than physiologic replacement doses; ocular steroid use is acceptable; (a) concomitant palliative radiation for the purposes of symptom management is allowed
* Women of childbearing potential (WOCBP) who: (a) are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for up to 26 weeks after cessation of study drug, or (b) have a positive pregnancy test at baseline, or (c) are pregnant or breastfeeding
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-11-29 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2024-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sapna Patel, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Pelster MS, Gruschkus SK, Bassett R, Gombos DS, Shephard M, Posada L, Glover MS, Simien R, Diab A, Hwu P, Carter BW, Patel SP. Nivolumab and Ipilimumab in Metastatic Uveal Melanoma: Results From a Single-Arm Phase II Study. J Clin Oncol. 2021 Feb 20;39(6):599-607. doi: 10.1200/JCO.20.00605. Epub 2020 Oct 30. PMID 33125309
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The accrual goal and dates were updated to match the new statistical design 10/2017.The enrollment changed to 39 participants. A total of 67 participants signed consent, 39 participants entered the study to participate in the trial in its current form w/combination metastatic therapy. 28 patients entered the study in its previous form when it was an adjuvant trial and then subsequently a monotherapy metastatic trial, and they are inevaluable for reporting results of the study in its current form
Groups:
- Treatment (Nivolumab, Ipilimumab): INDUCTION PHASE: Patients receive nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes during weeks 1, 4, 7, and 10. Treatment continues for 12 weeks in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Patients not experiencing disease progression or unacceptable toxicity by week 12 of the induction phase receive nivolumab IV every 2 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Ipilimumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV
Period: Overall Study
Arm/Group | Treatment (Nivolumab, Ipilimumab)
Started | 39
Completed | 35
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 2
Not completed — Lack of insurance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nivolumab, Ipilimumab)
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate, Defined Per RECIST 1.1
Description: RECIST 1.1 response is defined as >=30% reduction in sum of the longest diameter of target lesions
Time Frame: Up to 2 years of treatment plus 60 days from last study dose
Population: 5 patients not analyzed due to lack of follow-up efficacy imaging
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nivolumab, Ipilimumab)
Number analyzed (Participants) | 35
Participants
  Complete Response | 1
  Partial Response | 5
  Stable Disease | 11
  Progressive Disease | 16
  Unknown | 2

2. Secondary Outcome: Progression-Free Survival
Description: Time from enrollment to progressive disease or death. Progressive disease is defined per RECIST 1.1 as >=20% increase in the sum of the longest diameter of target lesions from nadir, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From date of enrollment until the date of progressive disease or date of death from any cause, whichever came first, and assessed up to 60 days after completion of study treatment, a median of 13.0 months
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Treatment (Nivolumab, Ipilimumab)
Number analyzed (Participants) | 35
Weeks | 5.5 [3.4 to 9.5]

3. Secondary Outcome: Overall Survival
Description: Measured from time of enrollment to death
Time Frame: From date of enrollment until the date of death from any cause, a median of 13.0 months
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Treatment (Nivolumab, Ipilimumab)
Number analyzed (Participants) | 35
Weeks | 19.1 [9.6 to NA] — The upper limit 95% Confidence Interval on Secondary Outcome Overall Survival as not enough "events" (deaths) have occurred past the median to calculate this upper limit of measure of dispersion.

4. Secondary Outcome: 1-year Overall Survival
Description: Measured as percentage of patients alive at 1 year from enrollment
Time Frame: Baseline up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nivolumab, Ipilimumab)
Number analyzed (Participants) | 35
Participants | 19

ADVERSE EVENTS:
Time Frame: From baseline to 60 days after last dose of study drug, a median of 13.0 months
Description: From baseline to 60 days after last dose of drug, a median of 13.0 months
Arm/Group | Treatment (Nivolumab, Ipilimumab)
All-Cause Mortality (participants affected / at risk) | 16/35
Serious Adverse Events (participants affected / at risk) | 2/35
Other Adverse Events (participants affected / at risk) | 32/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab, Ipilimumab) (N=35)
Death (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Nivolumab, Ipilimumab) (N=35)
Diarrhea (Gastrointestinal disorders) | 21
Increased ALT (Hepatobiliary disorders) | 17
Increased AST (Hepatobiliary disorders) | 14
Pruritus (Skin and subcutaneous tissue disorders) | 14
Hypothyroidism (Endocrine disorders) | 13
Rash (Skin and subcutaneous tissue disorders) | 11
Pyrexia (General disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Adrenal insufficiency (Endocrine disorders) | 4
Eye disorder (Eye disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT01585194/Prot_SAP_000.pdf